CLINICAL TRIAL: NCT00379483
Title: Extension Study of Iron Chelation Therapy With Deferasirox in Patients With Transfusional Iron Overload
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0105E1
Record Dates: First submitted 2005-10-14; First posted 2006-09-22 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Transfusional Iron Overload
Keywords: Transfusional iron overload; Deferasirox
MeSH Terms: interventions — Deferasirox

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: ICL670

SUMMARY:
A 1-year randomized Phase IIa core trial followed by a prolongation of 5 to 9 months was conducted to investigate the efficacy and safety of deferasirox in patients aged ≥ 18 years with transfusion-dependent iron overload.

The objective of this extension study is to assess the long-term safety of deferasirox and to provide treatment in patients with transfusional iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transfusional iron overload who have successfully completed the one year chelation treatment in the deferasirox trial or the food-effect sub-study and who were considered by the investigator eligible to continue chelation therapy with deferasirox

Exclusion Criteria:

* Pregnant or breast feeding patients
* Patients being considered by the investigator potentially unreliable and/or a history of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-07; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability of ICL670, at 3, 4, and 5 years treatment | at 3, 4, 5 years

SECONDARY OUTCOMES:
Change in liver iron content measured by SQUID, at 3, 4, and 5 years | at 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Italy (4):
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Torino